CLINICAL TRIAL: NCT02667717
Title: Efficacy and Safety of a Learning Program of Self- Rehabilitation Exercises by Mirror Therapy in the Complex Regional Pain Syndrome of the Upper Limb : a Multicentric Randomized Open Study.
Brief Title: Efficacy and Safety of a Learning Program of Self- Rehabilitation Exercises by Mirror Therapy
Acronym: AlgoMIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in including patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1508193; 2016-A00088-43 (Other: ANSM)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Reflex Sympathetic Dystrophy; Causalgia
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Causalgia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : Mirror Therapy (Experimental): Experimental group will perform mirror therapies during 16 weeks, added to the usual care. Therapy mirror sessions will take place at hospital units but also at home.
  Interventions: Behavioral: Mirror therapy; Behavioral: Usual care
- Control group : Usual care (Active Comparator): The control group will benefit from the usual care during 16 weeks. No mirror therapies will be performed to this group.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mirror therapy — The intervention is a mirror therapy. The mirror therapy consists in performing some movements with a mirror, the hand that is painful is hidden and the image of the healthy hand is reflected in the mirror. Patients looking at this image seems to see their painful hand moving.
  Arms: Experimental group : Mirror Therapy
Behavioral: Usual care — Patients will have the usual care as an intervention.

SUMMARY:
AlgoMIR project born thanks to a meeting between pain professionals and re-education staff. The goal of this project is to develop and evaluate a program of learning with exercises by mirror therapy, that could be easily shared with paramedic teams and easily adapted to different handicaps.

Researchers have chosen to select patients with re-education of the upper extremity to benefit from rehabilitation sessions either from physiotherapists present in their city, or of functional rehabilitation hospital units.

DETAILED DESCRIPTION:
The Complex Regional Painful Syndromes (CRPS) called in the past aglodystrophia, are characterized by the apparition of pain abnormally spread and intensive compared to the initial causal factor. They are usually associated to negligence of the painful limb, and avoidance movements that require care in rehabilitation that it is carried out in the physiotherapist center or functional rehabilitation unit at hospital.

Recently, mirror therapy has been proposed to correct dysfunctions : patients have to realize a movement with their two hands, observing the reflect of their healthy hand in a mirror, while their painful hand is hidden behind the mirror. After a learning phase, patients have to continue this kind of therapy independently.

AlgoMIR project born thanks to a meeting between pain professionals and re-education staff. The goal of this project is to develop and evaluate a program of learning with exercises by mirror therapy, that could be easily shared with paramedic teams and easily adapted to different handicaps.

Researchers have chosen to select patients with re-education of the upper extremity to benefit from rehabilitation sessions either from physiotherapists present in their city, or of functional rehabilitation hospital units.

The primary outcome of this project is to compare analgesic effect at 8 and 16 weeks of a therapy mirror re-education program associated to a usual care (M+R), and of a usual care program (R).

A second goal is to understand eventual difficulties met by the patients and improve efficacy of the autonomous becoming of patients using mirror therapy.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to Social Security
* CRPS (complex regional pain syndrome) type I or II defined by the criteria of Bruehl (Table 1)
* CRPS of the upper limb including the wrist and / or hand
* CRPS post-surgical or post-traumatic
* Average pain in the last 24 hours of intensity > = 30/100 on EVA (0 no pain, 100: worst pain imaginable )
* Evolution for over 3 months and less than 2 years
* Patients taking a stable background therapy for 15 days and not having received the following treatments in the previous months : bisphosphonate cure, infiltration, Qutenza, ketamine infusions
* Patients accepting a rehabilitation (physiotherapists or hospital units for patients included on Saint-Etienne and hospital units for patients included in Lyon and Saint- Vallier)

Exclusion Criteria:

* CRPS post stroke or drug
* Adhesive capsulitis isolated
* Cognitive or language difficulties preventing understanding instructions and / or a correct clinical evaluation
* Patient who already received a rehabilitation program with the use of mirror therapy or other virtual reality technology
* CRPS in connection with an accident caused by a third party for which a legal procedure is underway
* Major Depressive Episode
* Dissociative Disorders
* Visually impaired patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Compare the Visual Analogue Scale (EVA) of pain | Week 8
  Compare after 8 weeks the score of EVA of pain in the last 24 hours for patients who performed during 8 weeks :
  * a program of mirror therapy associated with the usual care (M+R) or
  * the usual care without mirror therapy

CONTACTS AND LOCATIONS:
Overall Officials: CREAC'H Christelle, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - MPR des Massues, Lyon
  - Centre médical de l'Argentière, Saint-Etienne
  - Chu Saint Etienne, Saint-Etienne
  - Consultation Douleur de la Mutualité de la Loire, Saint-Etienne
  - MPR de l'Hôpital Drôme Nord, Saint-Vallier

IPD SHARING:
Plan to Share IPD: No